CLINICAL TRIAL: NCT00623623
Title: STREAM (Strategic Reperfusion Early After Myocardial Infarction). Comparison of the Efficacy and Safety of a Strategy of Early Fibrinolytic Treatment With Tenecteplase and Additional Antiplatelet and Antithrombin Therapy Followed by Catheterisation Within 6-24 Hours or Rescue Coronary Intervention Versus a Strategy of Standard Primary PCI in Patients With Acute Myocardial Infarction Within 3 Hours of Onset of Symptoms
Brief Title: STREAM-Strategic Reperfusion (With Tenecteplase and Antithrombotic Treatment) Early After Myocardial Infarction
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1123.28; 2007-001219-44 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-02-15; First posted 2008-02-26 (Estimated); Results first posted 2019-08-01 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2019-06

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction | interventions — Enoxaparin; Catheterization; Tenecteplase; Clopidogrel

ARMS (2):
- Tenecteplase (Experimental): Early tenecteplase, clopidogrel and enoxaparin followed by routine or rescue coronary intervention
  Interventions: Drug: enoxaparin; Procedure: catheterisation; Drug: tenecteplase; Drug: clopidogrel
- primary PCI (Other): Standard primary PCI
  Interventions: Procedure: primary PCI

INTERVENTIONS:
Procedure: primary PCI — Standard primary PCI
  Arms: primary PCI
Drug: enoxaparin — Adjunctive treatment
  Arms: Tenecteplase
Procedure: catheterisation — Routine or rescue coronary intervention
  Arms: Tenecteplase
Drug: tenecteplase — Single, weight-adjusted i.v. bolus of tenecteplase
  Arms: Tenecteplase
Drug: clopidogrel — Adjunctive treatment
  Arms: Tenecteplase

SUMMARY:
This study aims at evaluating, in a proof of concept approach, the outcome of patients presenting with acute ST-elevation myocardial infarction within 3 hours of symptom onset in either a pre-hospital setting or community hospital emergency room without a PCI facility. Following randomisation a strategy of early tenecteplase and additional antiplatelet and antithrombin therapy followed by catheterisation within 6-24 hours with timely coronary intervention as appropriate (or by rescue coronary intervention if required) in Group A will be compared to primary PCI performed according to local standards in Group B.

The study is exploratory in nature and will examine this medical question. The efficacy and safety endpoints as well as mixed (efficacy and safety) composite endpoints up to or before 30 days following randomisation will be evaluated.

All clinical endpoints of main interest will be assessed as single or composite endpoints for evaluation of the trial objective. All statistical tests are of exploratory nature based on descriptive p-values for formal statistical hypotheses generation.

ELIGIBILITY:
Inclusion criteria:

1. Age equal or greater than 18 years
2. Onset of symptoms < 3 hours prior to randomisation 3.12-lead ECG indicative of an acute STEMI

4.Informed consent received

Exclusion criteria:

Medical history, procedures, medication administration or the presence of factors that would in general predispose to bleeding events and/or the inability to evaluate the study primary endpoint

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1899 (Actual)
Dates: Start 2008-03-01 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2012-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (201):
- Austria (9):
  - 1123.28.43009 Boehringer Ingelheim Investigational Site, Salzburg
  - 1123.28.43010 Boehringer Ingelheim Investigational Site, Salzburg
  - 1123.28.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43002 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43003 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43004 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43005 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43007 Boehringer Ingelheim Investigational Site, Vienna
  - 1123.28.43008 Boehringer Ingelheim Investigational Site, Vienna
- Belgium (4):
  - 1123.28.32060 Boehringer Ingelheim Investigational Site, Bornem
  - 1123.28.32010 Boehringer Ingelheim Investigational Site, Brussels
  - 1123.28.32070 Boehringer Ingelheim Investigational Site, Herentals
  - 1123.28.32040 Boehringer Ingelheim Investigational Site, Liège
- Brazil (11):
  - 1123.28.55010 Boehringer Ingelheim Investigational Site, Brasília
  - 1123.28.55020 Boehringer Ingelheim Investigational Site, Brasília
  - 1123.28.55008 Boehringer Ingelheim Investigational Site, Cabo Frio
  - 1123.28.55017 Boehringer Ingelheim Investigational Site, Campinas
  - 1123.28.55007 Boehringer Ingelheim Investigational Site, Porto Alegre
  - 1123.28.55001 Boehringer Ingelheim Investigational Site, Recife
  - 1123.28.55018 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1123.28.55028 Boehringer Ingelheim Investigational Site, Rio de Janeiro
  - 1123.28.55016 Boehringer Ingelheim Investigational Site, Sao Lourenço Do Sul
  - 1123.28.55004 Boehringer Ingelheim Investigational Site, São Paulo
  - 1123.28.55014 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (3):
  - 1123.28.11006 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1123.28.11505 Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - 1123.28.11002 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
- Chile (6):
  - 1123.28.13001 Boehringer Ingelheim Investigational Site, Santiago
  - 1123.28.13002 Boehringer Ingelheim Investigational Site, Santiago
  - 1123.28.13003 Boehringer Ingelheim Investigational Site, Santiago
  - 1123.28.13004 Boehringer Ingelheim Investigational Site, Santiago
  - 1123.28.13005 Boehringer Ingelheim Investigational Site, Santiago
  - 1123.28.13006 Boehringer Ingelheim Investigational Site, Santiago
- France (87):
  - 1123.28.3376A Boehringer Ingelheim Investigational Site, Ambérieu-en-Bugey
  - 1123.28.3329A Boehringer Ingelheim Investigational Site, Aubervilliers
  - 1123.28.3329B Boehringer Ingelheim Investigational Site, Aubervilliers
  - 1123.28.3329C Boehringer Ingelheim Investigational Site, Aubervilliers
  - 1123.28.3315A Boehringer Ingelheim Investigational Site, Besançon
  - 1123.28.3315B Boehringer Ingelheim Investigational Site, Besançon
  - 1123.28.3351A Boehringer Ingelheim Investigational Site, Besançon
  - 1123.28.3351B Boehringer Ingelheim Investigational Site, Besançon
  - 1123.28.3302A Boehringer Ingelheim Investigational Site, Bobigny
  - 1123.28.3302B Boehringer Ingelheim Investigational Site, Bobigny
  - 1123.28.3319A Boehringer Ingelheim Investigational Site, Bordeaux
  - 1123.28.3319B Boehringer Ingelheim Investigational Site, Bordeaux
  - 1123.28.3319C Boehringer Ingelheim Investigational Site, Bordeaux
  - 1123.28.3374A Boehringer Ingelheim Investigational Site, Bourg-en-Bresse
  - 1123.28.3383A Boehringer Ingelheim Investigational Site, Bourg-en-Bresse
  - 1123.28.3385A Boehringer Ingelheim Investigational Site, Bourg-en-Bresse
  - 1123.28.3347A Boehringer Ingelheim Investigational Site, Bourges
  - 1123.28.3347B Boehringer Ingelheim Investigational Site, Bourges
  - 1123.28.3347C Boehringer Ingelheim Investigational Site, Bourges
  - 1123.28.3355A Boehringer Ingelheim Investigational Site, Bron
  - 1123.28.3355B Boehringer Ingelheim Investigational Site, Bron
  - 1123.28.3382A Boehringer Ingelheim Investigational Site, Caluire-et-Cuire
  - 1123.28.3311A Boehringer Ingelheim Investigational Site, Châteauroux
  - 1123.28.3311B Boehringer Ingelheim Investigational Site, Châteauroux
  - 1123.28.3346A Boehringer Ingelheim Investigational Site, Châteauroux
  - 1123.28.3346B Boehringer Ingelheim Investigational Site, Châteauroux
  - 1123.28.3303A Boehringer Ingelheim Investigational Site, Clichy
  - 1123.28.3309A Boehringer Ingelheim Investigational Site, Dreux
  - 1123.28.3342A Boehringer Ingelheim Investigational Site, Dreux
  - 1123.28.3337A Boehringer Ingelheim Investigational Site, Évecquemont
  - 1123.28.3387A Boehringer Ingelheim Investigational Site, Fort de France Cedex
  - 1123.28.3388A Boehringer Ingelheim Investigational Site, Fort de France Cedex
  - 1123.28.3353A Boehringer Ingelheim Investigational Site, Grenoble
  - 1123.28.3353B Boehringer Ingelheim Investigational Site, Grenoble
  - 1123.28.3317A Boehringer Ingelheim Investigational Site, La Tronche
  - 1123.28.3317B Boehringer Ingelheim Investigational Site, La Tronche
  - 1123.28.3307A Boehringer Ingelheim Investigational Site, Le Chesnay
  - 1123.28.3339A Boehringer Ingelheim Investigational Site, Le Chesnay
  - 1123.28.3339B Boehringer Ingelheim Investigational Site, Le Chesnay
  - 1123.28.3336A Boehringer Ingelheim Investigational Site, Le Port-Marly
  - 1123.28.3301A Boehringer Ingelheim Investigational Site, Lille
  - 1123.28.3301B Boehringer Ingelheim Investigational Site, Lille
  - 1123.28.3325A Boehringer Ingelheim Investigational Site, Lille
  - 1123.28.3325B Boehringer Ingelheim Investigational Site, Lille
  - 1123.28.3326A Boehringer Ingelheim Investigational Site, Lille
  - 1123.28.3318A Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3318B Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3318C Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3356A Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3356B Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3369A Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3369B Boehringer Ingelheim Investigational Site, Lyon
  - 1123.28.3308A Boehringer Ingelheim Investigational Site, Melun
  - 1123.28.3308B Boehringer Ingelheim Investigational Site, Melun
  - 1123.28.3340A Boehringer Ingelheim Investigational Site, Melun
  - 1123.28.3340B Boehringer Ingelheim Investigational Site, Melun
  - 1123.28.3379A Boehringer Ingelheim Investigational Site, Montélimar
  - 1123.28.3328A Boehringer Ingelheim Investigational Site, Montfermeil
  - 1123.28.3328B Boehringer Ingelheim Investigational Site, Montfermeil
  - 1123.28.3328C Boehringer Ingelheim Investigational Site, Montfermeil
  - 1123.28.3313A Boehringer Ingelheim Investigational Site, Nantes
  - 1123.28.3313B Boehringer Ingelheim Investigational Site, Nantes
  - 1123.28.3349A Boehringer Ingelheim Investigational Site, Nantes
  - 1123.28.3349B Boehringer Ingelheim Investigational Site, Nantes
  - 1123.28.3322A Boehringer Ingelheim Investigational Site, Nice
  - 1123.28.3322B Boehringer Ingelheim Investigational Site, Nice
  - 1123.28.3322C Boehringer Ingelheim Investigational Site, Nice
  - 1123.28.3366A Boehringer Ingelheim Investigational Site, Nice
  - 1123.28.3375A Boehringer Ingelheim Investigational Site, Oyonnax
  - 1123.28.3331A Boehringer Ingelheim Investigational Site, Paris
  - 1123.28.3334A Boehringer Ingelheim Investigational Site, Paris
  - 1123.28.3371A Boehringer Ingelheim Investigational Site, Paris
  - 1123.28.3357A Boehringer Ingelheim Investigational Site, Pessac
  - 1123.28.3338A Boehringer Ingelheim Investigational Site, Poissy
  - 1123.28.3316A Boehringer Ingelheim Investigational Site, Pringy
  - 1123.28.3352A Boehringer Ingelheim Investigational Site, Pringy
  - 1123.28.3341A Boehringer Ingelheim Investigational Site, Quincy-sous-Sénart
  - 1123.28.3378A Boehringer Ingelheim Investigational Site, Romans-sur-Isère
  - 1123.28.3310A Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3310B Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3344A Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3345A Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3345B Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3345C Boehringer Ingelheim Investigational Site, Rouen
  - 1123.28.3377A Boehringer Ingelheim Investigational Site, Valence
  - 1123.28.3384A Boehringer Ingelheim Investigational Site, Valence
  - 1123.28.3373A Boehringer Ingelheim Investigational Site, Vienne
- Germany (6):
  - 1123.28.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1123.28.49006 Boehringer Ingelheim Investigational Site, Berlin
  - 1123.28.49008 Boehringer Ingelheim Investigational Site, Dortmund
  - 1123.28.49012 Boehringer Ingelheim Investigational Site, Duisburg
  - 1123.28.49052 Boehringer Ingelheim Investigational Site, Frankenthal
  - 1123.28.49026 Boehringer Ingelheim Investigational Site, Sömmerda
- Greece (11):
  - 1123.28.30012 Boehringer Ingelheim Investigational Site, Alexandroupoli
  - 1123.28.30001 Boehringer Ingelheim Investigational Site, Athens
  - 1123.28.30003 Boehringer Ingelheim Investigational Site, Chalikida
  - 1123.28.30006 Boehringer Ingelheim Investigational Site, Corinth
  - 1123.28.30011 Boehringer Ingelheim Investigational Site, Katerini
  - 1123.28.30014 Boehringer Ingelheim Investigational Site, Kavala
  - 1123.28.30002 Boehringer Ingelheim Investigational Site, Livadeia
  - 1123.28.30005 Boehringer Ingelheim Investigational Site, Thebes
  - 1123.28.30007 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1123.28.30010 Boehringer Ingelheim Investigational Site, Thessaloniki
  - 1123.28.30009 Boehringer Ingelheim Investigational Site, Véroia
- Italy (12):
  - 1123.28.39201 Boehringer Ingelheim Investigational Site, Ferrara
  - 1123.28.39002A Boehringer Ingelheim Investigational Site, Genova
  - 1123.28.39022 Boehringer Ingelheim Investigational Site, Genova
  - 1123.28.39004A Boehringer Ingelheim Investigational Site, Imperia
  - 1123.28.39200A Boehringer Ingelheim Investigational Site, Lagosanto (FE)
  - 1123.28.39001A Boehringer Ingelheim Investigational Site, Monza
  - 1123.28.39011 Boehringer Ingelheim Investigational Site, Monza
  - 1123.28.39082 Boehringer Ingelheim Investigational Site, Pescia (Pistoia)
  - 1123.28.39083 Boehringer Ingelheim Investigational Site, Pescia (Pistoia)
  - 1123.28.39008A Boehringer Ingelheim Investigational Site, Pistoia
  - 1123.28.39081 Boehringer Ingelheim Investigational Site, Pistoia
  - 1123.28.39041 Boehringer Ingelheim Investigational Site, Sanremo (IM)
- Norway (3):
  - 1123.28.47005 Boehringer Ingelheim Investigational Site, Hamar
  - 1123.28.47001 Boehringer Ingelheim Investigational Site, Oslo
  - 1123.28.47002 Boehringer Ingelheim Investigational Site, Oslo
- Peru (2):
  - 1123.28.19001 Boehringer Ingelheim Investigational Site, Lima
  - 1123.28.19004 Boehringer Ingelheim Investigational Site, Lima
- Poland (4):
  - 1123.28.48002 Boehringer Ingelheim Investigational Site, Gniezno
  - 1123.28.48006 Boehringer Ingelheim Investigational Site, Gniezno
  - 1123.28.48009 Boehringer Ingelheim Investigational Site, Grodzisk Wielopolski
  - 1123.28.48001 Boehringer Ingelheim Investigational Site, Poznan
- Russia (17):
  - 1123.28.70005 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1123.28.77005 Boehringer Ingelheim Investigational Site, Chelyabinsk
  - 1123.28.70009 Boehringer Ingelheim Investigational Site, Irkutsk
  - 1123.28.77009 Boehringer Ingelheim Investigational Site, Irkutsk
  - 1123.28.70002 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1123.28.77002 Boehringer Ingelheim Investigational Site, Kemerovo
  - 1123.28.70008 Boehringer Ingelheim Investigational Site, Murmansk
  - 1123.28.77008 Boehringer Ingelheim Investigational Site, Murmansk
  - 1123.28.77003 Boehringer Ingelheim Investigational Site, Nizhny Novgorod
  - 1123.28.70003 Boehringer Ingelheim Investigational Site, Nizhnyi Novgorod
  - 1123.28.70006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1123.28.70007 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1123.28.77006 Boehringer Ingelheim Investigational Site, Saint Petersburg
  - 1123.28.70004 Boehringer Ingelheim Investigational Site, Tomsk
  - 1123.28.77004 Boehringer Ingelheim Investigational Site, Tomsk
  - 1123.28.70001 Boehringer Ingelheim Investigational Site, Yekaterinburg
  - 1123.28.77001 Boehringer Ingelheim Investigational Site, Yekaterinburg
- Serbia (11):
  - 1123.28.38101 Boehringer Ingelheim Investigational Site, Belgrade
  - 1123.28.38103 Boehringer Ingelheim Investigational Site, Belgrade
  - 1123.28.38104 Boehringer Ingelheim Investigational Site, Belgrade
  - 1123.28.38106 Boehringer Ingelheim Investigational Site, Niš
  - 1123.28.38107 Boehringer Ingelheim Investigational Site, Niš
  - 1123.28.38108 Boehringer Ingelheim Investigational Site, Smederevo
  - 1123.28.38109 Boehringer Ingelheim Investigational Site, Šabac
  - 1123.28.38110 Boehringer Ingelheim Investigational Site, Vršac
  - 1123.28.38111 Boehringer Ingelheim Investigational Site, Zaječar
  - 1123.28.38104 Boehringer Ingelheim Investigational Site, Zemun
  - 1123.28.38105 Boehringer Ingelheim Investigational Site, Zemun
- Spain (6):
  - 1123.28.34001 Boehringer Ingelheim Investigational Site, Almería
  - 1123.28.34004 Boehringer Ingelheim Investigational Site, Granada
  - 1123.28.34003 Boehringer Ingelheim Investigational Site, Huelva
  - 1123.28.34007 Boehringer Ingelheim Investigational Site, Madrid
  - 1123.28.34002 Boehringer Ingelheim Investigational Site, Málaga
  - 1123.28.34011 Boehringer Ingelheim Investigational Site, Salamanca
- United Kingdom (9):
  - 1123.28.44600 Boehringer Ingelheim Investigational Site, Belfast
  - 1123.28.44610 Boehringer Ingelheim Investigational Site, Belfast
  - 1123.28.44210 Boehringer Ingelheim Investigational Site, Bristol
  - 1123.28.44220 Boehringer Ingelheim Investigational Site, Bristol
  - 1123.28.44200 Boehringer Ingelheim Investigational Site, Chippenham
  - 1123.28.44620 Boehringer Ingelheim Investigational Site, Dundonald
  - 1123.28.44110 Boehringer Ingelheim Investigational Site, Leicester
  - 1123.28.44630 Boehringer Ingelheim Investigational Site, Newry
  - 1123.28.44100 Boehringer Ingelheim Investigational Site, Nottingham

REFERENCES:
- [Derived] Armstrong PW, Zheng Y, Welsh RC, Sinnaeve PR, de Werf FV, Westerhout CM, Bainey KR. Primary Percutaneous Coronary Intervention within the First Hour: Insights from Early-Treated Patients with ST-Elevation Myocardial Infarction. Am Heart J. 2026 Jan 29:107363. doi: 10.1016/j.ahj.2026.107363. Online ahead of print. PMID 41619999
- [Derived] Bainey KR, Welsh RC, Zheng Y, Arias-Mendoza A, Ristic AD, Averkov OV, Lambert Y, Temple T, Ly E, Bogaerts K, Sinnaeve P, Westerhout CM, Van de Werf F, Armstrong PW; STREAM-2 Investigators. Pharmaco-invasive strategy and dosing of tenecteplase in STEMI patients 60 to <75 years: An inter-trial comparison of the STREAM-1 and STREAM-2 trials. Am Heart J. 2025 Jun;284:20-31. doi: 10.1016/j.ahj.2025.02.002. Epub 2025 Feb 12. PMID 39952376
- [Derived] Bainey KR, Welsh RC, Zheng Y, Arias-Mendoza A, Ristic AD, Averkov OV, Lambert Y, Kerr Saraiva JF, Sepulveda P, Rosell-Ortiz F, French JK, Music LB, Temple T, Ly E, Bogaerts K, Sinnaeve PR, Danays T, Westerhout CM, Van de Werf F, Armstrong PW; STREAM-2 Investigators. Pharmaco-Invasive Strategy With Half-Dose Tenecteplase in Patients With STEMI: Prespecified Pooled Analysis of Patients Aged >/=75 Years in STREAM-1 and 2. Circ Cardiovasc Interv. 2024 Dec;17(12):e014251. doi: 10.1161/CIRCINTERVENTIONS.124.014251. Epub 2024 Dec 17. PMID 39689189
- [Derived] Shavadia J, Welsh R, Gershlick A, Zheng Y, Huber K, Halvorsen S, Steg PG, Van de Werf F, Armstrong PW. Relationship Between Arterial Access and Outcomes in ST-Elevation Myocardial Infarction With a Pharmacoinvasive Versus Primary Percutaneous Coronary Intervention Strategy: Insights From the STrategic Reperfusion Early After Myocardial Infarction (STREAM) Study. J Am Heart Assoc. 2016 Jun 13;5(6):e003559. doi: 10.1161/JAHA.116.003559. PMID 28525886
- [Derived] Bainey KR, Fresco C, Zheng Y, Halvorsen S, Carvalho A, Ostojic M, Goldstein P, Gershlick AH, Westerhout CM, Van de Werf F, Armstrong PW; STREAM Investigators. Implications of ischaemic area at risk and mode of reperfusion in ST-elevation myocardial infarction. Heart. 2016 Apr;102(7):527-33. doi: 10.1136/heartjnl-2015-308075. Epub 2016 Jan 18. PMID 26783237
- [Derived] Shavadia J, Zheng Y, Dianati Maleki N, Huber K, Halvorsen S, Goldstein P, Gershlick AH, Wilcox R, Van de Werf F, Armstrong PW. Infarct Size, Shock, and Heart Failure: Does Reperfusion Strategy Matter in Early Presenting Patients With ST-Segment Elevation Myocardial Infarction? J Am Heart Assoc. 2015 Aug 24;4(8):e002049. doi: 10.1161/JAHA.115.002049. PMID 26304934
- [Derived] Gershlick AH, Westerhout CM, Armstrong PW, Huber K, Halvorsen S, Steg PG, Ostojic M, Goldstein P, Carvalho AC, Van de Werf F, Wilcox RG. Impact of a pharmacoinvasive strategy when delays to primary PCI are prolonged. Heart. 2015 May;101(9):692-8. doi: 10.1136/heartjnl-2014-306686. Epub 2015 Feb 17. PMID 25691510
- [Derived] Sinnaeve PR, Armstrong PW, Gershlick AH, Goldstein P, Wilcox R, Lambert Y, Danays T, Soulat L, Halvorsen S, Ortiz FR, Vandenberghe K, Regelin A, Bluhmki E, Bogaerts K, Van de Werf F; STREAM investigators. ST-segment-elevation myocardial infarction patients randomized to a pharmaco-invasive strategy or primary percutaneous coronary intervention: Strategic Reperfusion Early After Myocardial Infarction (STREAM) 1-year mortality follow-up. Circulation. 2014 Sep 30;130(14):1139-45. doi: 10.1161/CIRCULATIONAHA.114.009570. Epub 2014 Aug 26. PMID 25161043
- [Derived] Dianati Maleki N, Van de Werf F, Goldstein P, Adgey JA, Lambert Y, Sulimov V, Rosell-Ortiz F, Gershlick AH, Zheng Y, Westerhout CM, Armstrong PW. Aborted myocardial infarction in ST-elevation myocardial infarction: insights from the STrategic Reperfusion Early After Myocardial infarction trial. Heart. 2014 Oct;100(19):1543-9. doi: 10.1136/heartjnl-2014-306023. Epub 2014 Jun 10. PMID 24916050
- [Derived] Armstrong PW, Gershlick AH, Goldstein P, Wilcox R, Danays T, Lambert Y, Sulimov V, Rosell Ortiz F, Ostojic M, Welsh RC, Carvalho AC, Nanas J, Arntz HR, Halvorsen S, Huber K, Grajek S, Fresco C, Bluhmki E, Regelin A, Vandenberghe K, Bogaerts K, Van de Werf F; STREAM Investigative Team. Fibrinolysis or primary PCI in ST-segment elevation myocardial infarction. N Engl J Med. 2013 Apr 11;368(15):1379-87. doi: 10.1056/NEJMoa1301092. Epub 2013 Mar 10. PMID 23473396
- [Derived] Armstrong PW, Gershlick A, Goldstein P, Wilcox R, Danays T, Bluhmki E, Van de Werf F; STREAM Steering Committee. The Strategic Reperfusion Early After Myocardial Infarction (STREAM) study. Am Heart J. 2010 Jul;160(1):30-35.e1. doi: 10.1016/j.ahj.2010.04.007. PMID 20598969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, prospective, randomised, parallel, comparative international multicentre trial
Pre-assignment Details: All subjects were screened for eligibility to participate in trial. Subjects attended specialist sites to ensure that they (the subjects) met all implemented inclusion/exclusion criteria. Subjects were not to be randomised to trial drug if any of the specific entry criteria was violated.
Groups:
- Tenecteplase (Group A): Patients were administered Tenecteplase in a weight-adjusted dose regimen with clopidogrel (concomitant antiplatelet) and Enoxaparin (anticoagulant treatment) followed by timely coronary intervention (pharmacoinvasive treatment)
- Primary PCI (Group B): Patients received primary Percutaneous Coronary Intervention (PCI) according to local standards.
  Preceding and concomitant medication in particular antiplatelet and antithrombin drugs were to be given according to local standards and international guidelines.
Period: Overall Study
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Started | 950 | 949
Completed | 949 | 948
Not Completed | 1 | 1
Not completed — Previous enrolment into this study | 1 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All consented patients either randomised by Interactive Voice Response System (IVRS) or treated (i.e., manually allocated to treatment group) by the investigator. This population is also referred to as the intention-to-treat population (ITT).
Groups:
- Total: Total of all reporting groups
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B) | Total
Number analyzed (Participants) | 949 | 948 | 1897
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: FAS
  Years | 60 (12.42) | 60 (12.49) | 60 (12.46)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 195 | 208 | 403
    Male | 754 | 740 | 1494
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With All-cause Mortality, Cardiogenic Shock, Congestive Heart Failure and Recurrent Myocardial Infarction Within 30 Days for FAS.
Description: The number of observed patients with all-cause mortality, cardiogenic shock, congestive heart failure (CHF) and recurrent myocardial infarction within 30 days was reported for full analysis set (FAS).
Time Frame: 30 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 116 | 135
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); No confirmatory statistical hypothesis was pre-specified. All statistical tests were of exploratory nature based on descriptive p-values for formal statistical hypotheses generation; Test type: Other; p = 0.195, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 0.86, 95% CI 2-sided [0.68 to 1.08]

2. Secondary Outcome: Number of Patients With All Cause Mortality
Description: This is a key secondary endpoint. The number of observed patients with all cause mortality within 30 days was reported.
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 43 | 42
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.904, modified Poisson regression; modified Poisson regression model with robust error variance; Relative risk = 1.03, 95% CI 2-sided [0.68 to 1.55]

3. Secondary Outcome: Number of Patients With Cardiac Mortality
Description: This is a key secondary endpoint. The number of observed patients with cardiac mortality within 30 days was reported.
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 31 | 32
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.905, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 0.97, 95% CI 2-sided [0.60 to 1.58]

4. Secondary Outcome: Number of Patients With Cardiogenic Shock
Description: This is a key secondary endpoint. The number of observed patients with cardiogenic shock within 30 days was reported.
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 41 | 56
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.120, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 0.73, 95% CI 2-sided [0.49 to 1.08]

5. Secondary Outcome: Number of Patients With Congestive Heart Failure (CHF)
Description: This is a key secondary endpoint. The number of observed patients with congestive heart failure (CHF) within 30 days was reported.
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 57 | 72
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.170, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 0.79, 95% CI 2-sided [0.57 to 1.11]

6. Secondary Outcome: Number of Patients With Recurrent Myocardial Infarction (Reinfarction)
Description: This is a key secondary endpoint. The number of observed patients with recurrent myocardial infarction (reinfarction) within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 23 | 21
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.758, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 1.10, 95% CI 2-sided [0.61 to 1.97]

7. Secondary Outcome: Number of Patients With Rehospitalisation for Cardiac Reasons
Description: This is a key secondary endpoint. The number of observed patients with rehospitalisation for cardiac reasons within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 45 | 41
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.663, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 1.10, 95% CI 2-sided [0.73 to 1.66]

8. Secondary Outcome: Number of Patients With Rehospitalisation for Non-cardiac Reasons
Description: This is a key secondary endpoint. The number of observed patients with rehospitalisation for non-cardiac reasons within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 19 | 11
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.148, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 1.72, 95% CI 2-sided [0.82 to 3.60]

9. Secondary Outcome: Number of Patients With Serious Repeat Target Vessel Revascularization
Description: This is a key secondary endpoint. The number of observed patients with serious repeat target vessel revascularization within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 1 | 2
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.572, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 0.50, 95% CI 2-sided [0.05 to 5.52]

10. Secondary Outcome: Number of Patients With All Cause Death and Shock
Description: This is a key secondary endpoint. The number of observed patients with all cause death and shock within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 59 | 73
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.207, modified Poission Regression model; modified Poisson regression model with robust error variance; Relative risk = 0.81, 95% CI 2-sided [0.58 to 1.13]

11. Secondary Outcome: Number of Patients With All Cause Death and Shock and CHF
Description: This is a key secondary endpoint. The number of observed patients with all cause death and shock and CHF within 30 days was reported.
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 100 | 123
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.100, modified Poission Regression model; modified Poisson regression model with robust error variance; Relative risk = 0.81, 95% CI 2-sided [0.63 to 1.04]

12. Secondary Outcome: Number of Patients With All Cause Death and Shock and Reinfarction
Description: This is a key secondary endpoint. The number of observed patients with all cause death and shock and reinfarction within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 77 | 85
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.511, modified Poission Regression model; modified Poisson regression model with robust error variance; Relative Risk = 0.91, 95% CI 2-sided [0.67 to 1.22]

13. Secondary Outcome: Number of Patients With Total Fatal Stroke
Description: This is a key secondary endpoint. The number of observed patients with total fatal stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 7 | 4
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.369, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 1.75, 95% CI 2-sided [0.52 to 5.97]

14. Secondary Outcome: Number of Patients With Total Disabling Stroke
Description: This is a key secondary endpoint. The number of observed patients with total disabling stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 2 | 0
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.168, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 4.99, 95% CI 2-sided [0.51 to 49.08]

15. Secondary Outcome: Number of Patients With Total Non-disabling Stroke
Description: This is a key secondary endpoint. The number of observed patients with total non-disabling stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 8 | 1
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.049, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 8.02, 95% CI 2-sided [1.00 to 63.97]

16. Secondary Outcome: Number of Patients With Intracranial Haemorrhage
Description: This is a key secondary endpoint. The number of observed patients with intracranial haemorrhage within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 9 | 2
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.054, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 4.51, 95% CI 2-sided [0.98 to 20.82]

17. Secondary Outcome: Number of Patients With Ischaemic Stroke
Description: This is a key secondary endpoint. The number of observed patients with ischaemic stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 6 | 3
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.324, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 2.00, 95% CI 2-sided [0.50 to 7.99]

18. Secondary Outcome: Number of Patients With Total Stroke (All Types)
Description: This is a key secondary endpoint. The number of observed patients with total stroke (all types) within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 15 | 5
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.032, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 3.01, 95% CI 2-sided [1.10 to 8.24]

19. Secondary Outcome: Number of Patients With Major Non-intracranial Bleeds Including Blood Transfusions
Description: This is a key secondary endpoint. The number of observed patients with major non-intracranial bleeds including blood transfusions within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 61 | 45
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.111, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 1.36, 95% CI 2-sided [0.93 to 1.97]

20. Secondary Outcome: Number of Patients With Minor Non-intracranial Bleeds
Description: This is a key secondary endpoint. The number of observed patients with minor non-intracranial bleeds within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 206 | 191
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.397, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 1.08, 95% CI 2-sided [0.91 to 1.28]

21. Secondary Outcome: Number of Patients With Total Non-intracranial Bleeds
Description: This is a key secondary endpoint. The number of observed patients with total non-intracranial bleeds within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 267 | 236
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.107, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 1.13, 95% CI 2-sided [0.97 to 1.31]

22. Secondary Outcome: Number of Patients With Serious Resuscitated Ventricular Fibrillation
Description: This is a key secondary endpoint. The number of observed patients with serious resuscitated ventricular fibrillation within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 32 | 38
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.471, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 0.84, 95% CI 2-sided [0.53 to 1.34]

23. Secondary Outcome: Number of Patients With Serious Resuscitated Ventricular Fibrillation in Association With Invasive Procedures
Description: This is a key secondary endpoint. The number of observed patients with serious resuscitated ventricular fibrillation in association with invasive procedures (occurring at any time during catheterisation or urgent/elective PCI) within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 10 | 29
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 0.35, 95% CI 2-sided [0.17 to 0.71]

24. Secondary Outcome: Number of Patients With All Cause Death and Non-fatal Stroke
Description: This is a key secondary endpoint. The number of observed patients with all cause death and non-fatal stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 50 | 43
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); Test type: Other; p = 0.451, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative risk = 1.17, 95% CI 2-sided [0.78 to 1.73]

25. Secondary Outcome: Number of Patients With All Cause Death and Shock and CHF and Reinfarction and Disabling Stroke
Description: This is a key secondary endpoint. The number of observed patients with all cause death and shock and CHF and reinfarction and disabling stroke within 30 days was reported
Time Frame: 30 days
Population: FAS
Measure: Count of Participants; unit: Participants
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
Number analyzed (Participants) | 949 | 948
Participants | 117 | 135
Statistical Analysis 1: Comparison: Tenecteplase (Group A) vs Primary PCI (Group B); Test type: Other; p = 0.220, modified Poisson regression model; modified Poisson regression model with robust error variance; Relative Risk = 0.87, 95% CI 2-sided [0.69 to 1.09]

ADVERSE EVENTS:
Time Frame: From first drug administration until end of tiral, up to 30 days
Arm/Group | Tenecteplase (Group A) | Primary PCI (Group B)
All-Cause Mortality (participants affected / at risk) | 43/949 | 42/948
Serious Adverse Events (participants affected / at risk) | 146/949 | 164/948
Other Adverse Events (participants affected / at risk) | 0/949 | 0/948
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tenecteplase (Group A) (N=949) | Primary PCI (Group B) (N=948)
Accelerated idioventricular rhythm (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 0 | 1
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 4 | 11
Atrioventricular block (Cardiac disorders) | 9 | 14
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 3 | 4
Cardiac arrest (Cardiac disorders) | 10 | 16
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 2 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 2 | 0
Coronary artery occlusion (Cardiac disorders) | 3 | 8
Coronary artery perforation (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Coronary artery thrombosis (Cardiac disorders) | 1 | 1
Intracardiac thrombus (Cardiac disorders) | 2 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 3
Myocardial ischaemia (Cardiac disorders) | 5 | 2
Myocardial rupture (Cardiac disorders) | 5 | 1
Parasystole (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 4
Pericarditis (Cardiac disorders) | 9 | 7
Postinfarction angina (Cardiac disorders) | 2 | 0
Pulseless electrical activity (Cardiac disorders) | 5 | 3
Right ventricular failure (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Sinus arrhythmia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 41 | 46
Ventricular tachycardia (Cardiac disorders) | 11 | 13
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 4 | 4
Device occlusion (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 2 | 2
Necrosis (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Thrombosis in device (General disorders) | 3 | 4
Hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 1 | 0
Bronchopneumonia (Infections and infestations) | 0 | 1
Endocarditis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Mediastinitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 7 | 5
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 0
Septic shock (Infections and infestations) | 3 | 0
Sputum purulent (Infections and infestations) | 1 | 0
Toxic shock syndrome (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 0
Fat embolism (Injury, poisoning and procedural complications) | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood electrolytes abnormal (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 0 | 1
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Pulse absent (Investigations) | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuromyopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 2 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 3 | 4
Renal failure acute (Renal and urinary disorders) | 3 | 5
Renal impairment (Renal and urinary disorders) | 2 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 11 | 14
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cardiac pacemaker insertion (Surgical and medical procedures) | 1 | 0
Coronary revascularisation (Surgical and medical procedures) | 1 | 2
Mechanical ventilation (Surgical and medical procedures) | 1 | 0
Resuscitation (Surgical and medical procedures) | 0 | 1
Aortic dissection (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 4
Peripheral ischaemia (Vascular disorders) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.